CLINICAL TRIAL: NCT05168449
Title: The Impact of Pharmacist - Led Mobile Application on Medication Adherence and Efficacy in Chronic Kidney Disease Patients
Brief Title: The Impact of Pharmacist-led Mobile Application on Adherence in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaza Gamal Abdel Fattah Ali Mohamed, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CL (2871)
Record Dates: First submitted 2021-11-24; First posted 2021-12-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Adherence, Medication
MeSH Terms: conditions — Renal Insufficiency, Chronic; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group will be provided with usual care. Intervention group will be provided in addition to the usual care, with an access to the previously described mobile application
- Intervention Group (Experimental): Intervention group will be provided in addition to the usual care, with an access to the mobile application
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Application — mobile phone applications directed to chronic kidney disease patients to improve their medication.
  Arms: Intervention Group

SUMMARY:
The aim of the study is to assess the impact of pharmacist led mobile application on adherence and efficacy of medication in chronic kidney disease patients

DETAILED DESCRIPTION:
This is a prospective randomized two group pharmacist-led interventional study that will be conducted in a private nephrology clinic. The study will involve introduction of the mobile phone applications to chronic kidney disease patients to improve their adherence to the prescribed medications.

Recruited patients will be randomly divided in two groups; intervention group and control group, with baseline evaluation of outcomes to be measured.

Control group will be provided with usual care. Intervention group will be provided in addition to the usual care, with an access to the mobile application after a simple training for app usage. Both groups will be followed for a period of 3 months.

The study will include the development, validation and the testing for evaluating the specially designed mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Stages 2-5 of chronic kidney disease
* Literate
* Ownership of android smart phone compatible with the application
* Poly-pharmacy

Exclusion Criteria:

* On dialysis due to loss of kidney function
* Pregnancy due to altered physiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence | Change from baseline at 3 months
  Using a medication adherence questionnaire.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate/ creatinine clearance | Change from baseline at 3 months
  Calculated using serum creatinine lab results obtained from clinic.
Change in systolic and diastolic blood pressure | Change from baseline at 3 months
  To be measured in clinic.
Change in HbA1c | Change from baseline at 3 months
  Lab results obtained from clinic.
Change in mobile application usability and acceptability by patients | Change from baseline at 3 months
  Using System Usability Scale (SUS) questionnaire. (scale 0-100 with higher score meaning better usability)

CONTACTS AND LOCATIONS:
Overall Officials: Shaza Gamal, Bsc, Principal Investigator — Teaching Assistant
Locations (1):
- Private Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamal S, Elseasi AMA, Sabry NA, Farid SF. Impact of pharmacist led mobile application on medication adherence and efficacy in chronic kidney disease. NPJ Digit Med. 2025 May 30;8(1):325. doi: 10.1038/s41746-025-01742-8. PMID 40447835